CLINICAL TRIAL: NCT03263143
Title: Early Palliative Care in the Medical Intensive Care Unit
Brief Title: Palliative Care in the ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Marin Kollef, Professor, Division of Pulmonary and Critical Care Medicine, Washington University School of Medicine
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 201707067; NCT03210116 (obsolete NCT alias)
Record Dates: First submitted 2017-07-26; First posted 2017-08-28 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Palliative Care
MeSH Terms: interventions — Palliative Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention)
- Early Palliative Care Consultation (Other)
  Interventions: Other: Palliative Care

INTERVENTIONS:
Other: Palliative Care — Palliative Care Consultation within 24 to 48 hours after admission
  Arms: Early Palliative Care Consultation

SUMMARY:
The study compares early palliative care consultation to standard of care in the medical intensive care unit (ICU). The study will assess if the intervention leads to an increased proportion of clearly delineated goals of care and examine if this intervention leads to decreased healthcare resource utilization such as length of stay, duration of intensive treatments including mechanical ventilation, and hospital re-admissions.

DETAILED DESCRIPTION:
* The medical intensive care unit will be split into two groups, assigned as either early palliative care consultation or standard of care. Current standard of care in the ICU is that primary clinician providers determine the need and time for palliative care consultation, which can occur approximately 5 - 14 days after admission.
* A palliative care screening tool will be used to determine if a newly admitted patient is eligible for palliative care consultation.
* Up to two patients per ICU per weekday will be enrolled into the study, due to workload limitations on the palliative care consult team.
* For patients in the intervention group, a palliative care consultation will be performed within 48 hours of ICU admission and patients will be followed throughout their hospitalization.
* Patients in the standard of care group will receive usual care. Palliative care may be consulted at the primary team's clinical discretion.
* The two medical ICU groups will be crossed over after three months with a washout period of six weeks, for a total of approximately eight months of study
* Electronic medical records will be reviewed after patient discharge to collect data on clinical outcomes as described elsewhere

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the ICU in the last 24 hours
* Admitted from Skilled nursing facility (SNF), long term acute care (LTAC)facility, long term ventilator care (vent LTC) unit, or home care with private duty nursing with activity of daily living (ADL) dependencies
* End-stage dementia, amyotrophic lateral sclerosis, Parkinson's, multiple sclerosis
* Advanced or Metastatic Cancer
* Cardiac or respiratory arrest with neurological compromise
* Multi- organ system failure (more than 2 organ failures)
* Known diagnosis of end stage organ disease including cirrhosis, end-stage renal disease, congestive heart failure New York Heart Association >III, chronic obstructive pulmonary disease on home O2
* Shock requiring > 6 hours of vasopressors or inotropes
* Acute Respiratory failure requiring intubation or BiPAP
* Admitted to ICU with hospital length of stay of more than 5 days or ICU readmission with the same diagnosis in 30 days.

Exclusion Criteria:

* All stem cell transplant patients, for solid organ transplant, if undergoing evaluation for solid organ transplant or within 1 year post-transplant.
* Patients who do not speak English if interpreter is unavailable
* Patients without capacity to participate in palliative care discussions without a surrogate available
* Patients or patient surrogate refusal of palliative care consultation
* Prior Palliative Care Consultation during the same hospitalization
* For purposes of primary outcome analysis, patients determined to already be DNR/DNI at time of ICU admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2017-08-07 (Actual); Primary Completion 2018-06-09 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Change in code status to do-not-resuscitate/do-not-intubate | Through patient admission until discharge, charts reviewed an average of one month after discharge
  As determined by code status orders in the electronic medical record

SECONDARY OUTCOMES:
Number of participants with Cardiopulmonary Resuscitation (CPR) performed | Through study completion, an average of 6 months
Mechanical Ventilation usage and duration | After date of discharge, charts reviewed an average of one month after discharge
Hospital Length of Stay | After date of discharge, charts reviewed an average of one month after discharge
ICU Length of Stay | After date of discharge, charts reviewed an average of one month after discharge
In-hospital mortality | After date of discharge, charts reviewed an average of one month after discharge
  Excluding patients transitioned to hospice prior to death
30-day mortality | One to two months after patient discharge, verified at study completion
  Including all patients, including those on hospice
Hospice transition or discharge | Through patient admission until discharge, charts reviewed an average of one month after discharge
Post-discharge ER visits and/or readmissions | One to two months after patient discharge, verified at study completion
  Determined by review of the BJC healthcare system electronic medical record
Total hospital operating cost | Through study completion, an average of 6 months
Vasopressor usage and duration | After date of discharge, charts reviewed an average of one month after discharge
Antibiotic usage and duration | After date of discharge, charts reviewed an average of one month after discharge
Number of participants treated with hemodialysis | Through study completion, an average of six months
Number of participants with tracheostomy performed during hospital stay | Through study completion, an average of six months

CONTACTS AND LOCATIONS:
Locations (1):
- Barnes Jewish Hospital, St Louis, Missouri, United States

REFERENCES:
- [Background] Adelson K, Paris J, Horton JR, Hernandez-Tellez L, Ricks D, Morrison RS, Smith CB. Standardized Criteria for Palliative Care Consultation on a Solid Tumor Oncology Service Reduces Downstream Health Care Use. J Oncol Pract. 2017 May;13(5):e431-e440. doi: 10.1200/JOP.2016.016808. Epub 2017 Mar 17. PMID 28306372
- [Background] Aslakson R, Cheng J, Vollenweider D, Galusca D, Smith TJ, Pronovost PJ. Evidence-based palliative care in the intensive care unit: a systematic review of interventions. J Palliat Med. 2014 Feb;17(2):219-35. doi: 10.1089/jpm.2013.0409. PMID 24517300
- [Background] Hsu-Kim C, Friedman T, Gracely E, Gasperino J. Integrating Palliative Care into Critical Care: A Quality Improvement Study. J Intensive Care Med. 2015 Sep;30(6):358-64. doi: 10.1177/0885066614523923. Epub 2014 Mar 5. PMID 24603677
- [Background] Khandelwal N, Kross EK, Engelberg RA, Coe NB, Long AC, Curtis JR. Estimating the effect of palliative care interventions and advance care planning on ICU utilization: a systematic review. Crit Care Med. 2015 May;43(5):1102-11. doi: 10.1097/CCM.0000000000000852. PMID 25574794
- [Background] Kyeremanteng K, Gagnon LP, Thavorn K, Heyland D, D'Egidio G. The Impact of Palliative Care Consultation in the ICU on Length of Stay: A Systematic Review and Cost Evaluation. J Intensive Care Med. 2018 Jun;33(6):346-353. doi: 10.1177/0885066616664329. Epub 2016 Aug 31. PMID 27582396
- [Background] Penrod JD, Pronovost PJ, Livote EE, Puntillo KA, Walker AS, Wallenstein S, Mercado AF, Swoboda SM, Ilaoa D, Thompson DA, Nelson JE. Meeting standards of high-quality intensive care unit palliative care: clinical performance and predictors. Crit Care Med. 2012 Apr;40(4):1105-12. doi: 10.1097/CCM.0b013e3182374a50. PMID 22202706
- [Background] Mun E, Ceria-Ulep C, Umbarger L, Nakatsuka C. Trend of Decreased Length of Stay in the Intensive Care Unit (ICU) and in the Hospital with Palliative Care Integration into the ICU. Perm J. 2016 Fall;20(4):16-036. doi: 10.7812/TPP/16-036. Epub 2016 Aug 31. PMID 27644048
- [Background] Braus N, Campbell TC, Kwekkeboom KL, Ferguson S, Harvey C, Krupp AE, Lohmeier T, Repplinger MD, Westergaard RP, Jacobs EA, Roberts KF, Ehlenbach WJ. Prospective study of a proactive palliative care rounding intervention in a medical ICU. Intensive Care Med. 2016 Jan;42(1):54-62. doi: 10.1007/s00134-015-4098-1. Epub 2015 Nov 10. PMID 26556622
- [Derived] Ma J, Chi S, Buettner B, Pollard K, Muir M, Kolekar C, Al-Hammadi N, Chen L, Kollef M, Dans M. Early Palliative Care Consultation in the Medical ICU: A Cluster Randomized Crossover Trial. Crit Care Med. 2019 Dec;47(12):1707-1715. doi: 10.1097/CCM.0000000000004016. PMID 31609772